CLINICAL TRIAL: NCT06948175
Title: Abdominal Transcutaneous Electrical Stimulation to Alleviate Neurogenic Bowel Dysfunction in People With Chronic Spinal Cord Injury
Brief Title: Abdominal Electrical Stimulation for Bowel Dysfunction in SCI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Praxis Spinal Cord Institute (Other); Glenrose Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00150346; G2025-13 (Other Grant/Funding Number: Praxis Spinal Cord Institute)
Record Dates: First submitted 2025-04-08; First posted 2025-04-29 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Chronic Spinal Cord Injury
Keywords: spinal cord injury; functional electrical stimulation; transcutaneous electrical stimulation; neurogenic bowel dysfunction; bowel dysfunction; abdominal electrical stimulation; sensory stimulation; defecation time; bowel transit time; stool consistency; bowel routine
MeSH Terms: conditions — Spinal Cord Injuries; Intestinal Diseases

STUDY DESIGN:
Intervention Model Description: The study uses an interrupted time-series design with 4 phases of observation and 3 changes in condition in a single group of participants. The conditions per phase and phase durations are as follows:
  Phase 1 (duration 2 weeks): Participants apply their usual bowel routine for baseline observation.
  Phase 2 (duration 4 weeks): In case that the initial assessment resulted in recommendations for improvement to the participant's usual bowel routine (See 2. Interventions), participants apply their optimized bowel routine in Phase 2 for 4 weeks. If no bowel routine adjustment was recommended, Phase 2 is omitted.
  Phase 3 (duration 8 weeks): Participants apply abdominal TES for 30 minutes prior to every bowel routine. In case the bowel routine was optimized, they keep applying the optimized bowel routine.
  Phase 4 (duration 4 weeks): Participants go back to their optimized bowel routine only, without using abdominal TES.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abdominal TES (Experimental): Abdominal transcutaneuous electrical stimulation (TES)
  Interventions: Device: Abdominal transcutaneous electrical stimulation (TES)

INTERVENTIONS:
Device: Abdominal transcutaneous electrical stimulation (TES) — Low-intensity sensory abdominal transcutaneous electrical stimulation (TES)

SUMMARY:
Many people with spinal cord injury (SCI) have bowel problems resulting in constipation and need a long time to empty the bowel. Some people spend an hour or more to empty their bowel. The investigators want test if using a small device to deliver electrical pulses to the belly (abdomen), would improve bowel function. The investigators hope that electrical stimulation will shorten the time needed to evacuate the bowel (defecation), improve stool consistency, and speed up food passing through the bowel. A pilot study found that electrical stimulation of the belly can speed up defecation if stimulation is making the abdominal muscles contract and squeeze the belly, which is what the investigators expected. However, some results suggested that people may benefit from low stimulation levels without making the muscles contract.

Therefore, the investigators will do small study at the University of Alberta on 12 people who lived with SCI for more than 1 year, to find out the best way to apply the electrical stimulation, and to better understand how it works. The participants will use an electrical stimulator at home, to stimulate the skin with 4 sticky pads attached over the abdomen, without causing the muscles to contract. During a 2-month period, they will use the stimulator for 30 minutes before every bowel routine. The investigators will compare how long it takes to empty the bowel, stool consistency, and how long it takes for food to pass through the bowel, with and without using the electrical stimulator.

ELIGIBILITY:
Inclusion Criteria:

1. Traumatic or non-traumatic SCI
2. >1 year post injury
3. Injury level C2 - S5 (NLI, neurological level of injury)
4. AIS A, B, C, D (American Spinal Injury Association Impairment Scale)
5. Feels defecation takes too long and wants to do something about it
6. Defecation takes > 30 minutes

Exclusion Criteria:

1. Bladder stimulator
2. Inflammatory bowel disease
3. Pregnancy
4. Unable to give consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Mean defecation time at 2 weeks | 2 weeks after enrollment (after 2 weeks of usual bowel routine)
  Mean defecation time for all bowel routines from 0 to 2 weeks (2 weeks of usual bowel routine). Defecation time = time from initiation of bowel movement to the end of stool evacuation.
Mean defecation time at 6 weeks | 6 weeks after enrollment (after 4 weeks of optimized bowel routine)
  Mean defecation time for all bowel routines from 2 to 6 weeks (4 weeks of optimized bowel routine). Defecation time = time from initiation of bowel movement to the end of stool evacuation.
Mean defecation time at 14 weeks | 14 weeks after enrollment (after 8 weeks of abdominal TES)
  Mean defecation time for all bowel routines from 6 to 14 weeks (8 weeks of abdominal TES). Defecation time = time from initiation of bowel movement to the end of stool evacuation.
Mean defecation time at 18 weeks | 18 weeks after enrollment (after 4 weeks of usual bowel routine)
  Mean defecation time for all bowel routines from 14 to 18 weeks (4 weeks of usual bowel routine). Defecation time = time from initiation of bowel movement to the end of stool evacuation.

SECONDARY OUTCOMES:
Bristol Stool Form | Every bowel routine
  The Bristol Stool Form Scale will be used to score stool form or consistency. The scale from 1-7 is scored using a 1-page document with a graphic and description of 7 different types of stool
Bowel Transit Time at 2 weeks | 2 weeks after enrollment (after 2 weeks of usual bowel routine)
  Bowel transit time is defined as the time from ingestion of food to time of evacuation, and will be measured using the "corn test". The participants will eat a full can of corn, on its own or with a meal, and write down the date and time of ingestion on a log sheet. They will then inspect stool after every defecation for the presence of corn kernels, and write down the date and time of the first appearance of corn in the stool
Bowel Transit Time at 6 weeks | 6 weeks after enrollment (after 4 weeks of optimized bowel routine)
  Bowel transit time is defined as the time from ingestion of food to time of evacuation, and will be measured using the "corn test". The participants will eat a full can of corn, on its own or with a meal, and write down the date and time of ingestion on a log sheet. They will then inspect stool after every defecation for the presence of corn kernels, and write down the date and time of the first appearance of corn in the stool
Bowel Transit Time at 14 weeks | 14 weeks after enrollment (after 8 weeks of abdominal TES)
  Bowel transit time is defined as the time from ingestion of food to time of evacuation, and will be measured using the "corn test". The participants will eat a full can of corn, on its own or with a meal, and write down the date and time of ingestion on a log sheet. They will then inspect stool after every defecation for the presence of corn kernels, and write down the date and time of the first appearance of corn in the stool
Bowel Transit Time at 18 weeks | 18 weeks after enrollment (after 4 weeks of usual bowel routine)
  Bowel transit time is defined as the time from ingestion of food to time of evacuation, and will be measured using the "corn test". The participants will eat a full can of corn, on its own or with a meal, and write down the date and time of ingestion on a log sheet. They will then inspect stool after every defecation for the presence of corn kernels, and write down the date and time of the first appearance of corn in the stool
Neurogenic Bowel Dysfunction Score (NBDS) at 2 weeks | 2 weeks after enrollment (after 2 weeks of usual bowel routine)
  The Neurogenic Bowel Dysfunction Score is a score from 0 to 47 documenting severity of bowel dysfunction, and is based on a 1-page form with 10 questions about frequency and time used for defecation, medication use for constipation and incontinence, use of digital stimulation, fecal incontinence and flatus, peri-anal skin problems
Neurogenic Bowel Dysfunction Score (NBDS) at 6 weeks | 6 weeks after enrollment (after 4 weeks of optimized bowel routine)
  The Neurogenic Bowel Dysfunction Score is a score from 0 to 47 documenting severity of bowel dysfunction, and is based on a 1-page form with 10 questions about frequency and time used for defecation, medication use for constipation and incontinence, use of digital stimulation, fecal incontinence and flatus, peri-anal skin problems
Neurogenic Bowel Dysfunction Score (NBDS) at 14 weeks | 14 weeks after enrollment (after 8 weeks of abdominal TES)
  The Neurogenic Bowel Dysfunction Score is a score from 0 to 47 documenting severity of bowel dysfunction, and is based on a 1-page form with 10 questions about frequency and time used for defecation, medication use for constipation and incontinence, use of digital stimulation, fecal incontinence and flatus, peri-anal skin problems
Neurogenic Bowel Dysfunction Score (NBDS) at 18 weeks | 18 weeks after enrollment (after 4 weeks of usual bowel routine)
  The Neurogenic Bowel Dysfunction Score is a score from 0 to 47 documenting severity of bowel dysfunction, and is based on a 1-page form with 10 questions about frequency and time used for defecation, medication use for constipation and incontinence, use of digital stimulation, fecal incontinence and flatus, peri-anal skin problems
Participant Feedback | 18 weeks after enrollment (end of study)
  At the end of the study, the participants participate in a semi-structured interview (in person or over the phone) to evaluate their level of satisfaction and acceptability of abdominal TES, problems that were encountered, potential benefits they perceived

OTHER OUTCOMES:
ISNCSCI | Baseline
  A neurological assessment will be performed according to the International Standards for Neurological Classification of Spinal Cord Injury, in order to determine the ASIA Impairment Score (AIS) and neurological level of injury. The AIS score is based on manual testing of strength of 10 key muscle groups in upper and lower extremities, sensory response to light touch and pinprick at 28 key sensory points on each side of the whole body, and anal responses.
Demographics & medical history | Baseline
  Demographic information, past medical history, information on SCI and current medical issues

CONTACTS AND LOCATIONS:
Overall Officials: Chester Ho, MD, Principal Investigator — University of Alberta, Faculty of Medicine and Dentistry
Locations (1):
- Glenrose Rehabilitation Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided